CLINICAL TRIAL: NCT02953275
Title: Synergistic Effect of Vedolizumab and Pentoxifylline in the Management of Patients With Inflammatory Bowel Disease
Brief Title: Synergistic Effect of Vedolizumab and Pentoxifylline
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Amar Deshpande, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20160543
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab; Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- vedolizumab plus pentoxifylline (Experimental): Patients will receive standard induction and maintenance dosing of vedolizumab 300 mg intravenously as well as pentoxifylline 400 mg orally thrice daily.
  Interventions: Drug: vedolizumab; Drug: Pentoxifylline
- vedolizumab plus placebo (Placebo Comparator): Patients will receive standard induction and maintenance dosing of vedolizumab 300 mg intravenously as well as placebo orally thrice daily.
  Interventions: Drug: vedolizumab; Drug: placebo

INTERVENTIONS:
Drug: vedolizumab — standard of care
  Other Names: Entyvio
Drug: Pentoxifylline — added to vedolizumab
  Other Names: Trental
  Arms: vedolizumab plus pentoxifylline
Drug: placebo — added to vedolizumab
  Arms: vedolizumab plus placebo

SUMMARY:
The purpose of this study is to determine the synergistic effect and clinical benefits of vedolizumab and pentoxifylline in the management of patients with inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active Crohn's disease (CD) defined by blood lab values, stool markers, abnormal MR enterography imaging, or colonoscopic findings
* Patients who are good candidates to start standard dosing of vedolizumab
* Patients who have not used an off-label or investigational drug for CD in the 8 weeks prior to screening
* Patients who have met the washout period of 8 weeks for infliximab, 4 weeks for certolizumab pegol, and 2 weeks for adalimumab if there is a history of anti-TNF exposure and 8 weeks if there is a history of exposure to natalizumab
* Oral aminosalicylates are allowed during the study, provided that the dose has been stable for at least 2 weeks prior to screening
* Oral corticosteroids are allowed provided that the dose is prednisone ≤40 mg/day or equivalent and/or budesonide ≤9mg/day and has been stable for at least 2 weeks prior to screening
* Patients are able to discontinue thiopurines (azathioprine and 6-mercaptopurine) or methotrexate upon initiation of vedolizumab
* Rectal therapies, narcotics, anti-diarrheals, probiotics, and antibiotics will be permitted at investigator discretion

Exclusion Criteria:

* Contraindications or history of allergy to PTX
* Known interaction of PTX with patient's current medications
* Use of an off-label or investigational drug for CD in the 8 weeks prior to first VDZ infusion
* Pregnancy
* GFR <30 at any time in the 6 months prior to first infusion of VDZ
* Documented cirrhosis
* Age <18 or >80 years old
* Contraindication to colonoscopy at 24 week study time-point

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
proportion of patients in clinical remission | week 14

SECONDARY OUTCOMES:
number of new major and minor infections | week 24
number of episodes of nephrotoxicity | week 24
number of episodes of hepatotoxicity | week 24
number of episodes of myelosuppression | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Amar R Deshpande, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Crohn's and Colitis Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No